CLINICAL TRIAL: NCT07242924
Title: Enhanced Recovery After Emergency Cesarean Section: A Comparative Study Assessing Postoperative Recovery and Outcomes
Acronym: ERAS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Abbady Hussein, Resident physician, Assiut University
Other Study IDs: ERAS after emergency cs
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: ERAS; Cesarean Section Pain
Keywords: ERAS; ERAS, emergency cs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enhanced Recovery After Surgery protocol for emergency cesarean section: Application of ERAS protocol delivered perioperatively and postoperatively as per institutional ERAS guidelines.

SUMMARY:
Cesarean section (CS) remains one of the most common major surgical procedures worldwide, with emergency CS accounting for approximately 30% of cases. Emergency CS presents unique challenges including increased maternal stress, higher complication rates, and prolonged recovery compared to elective procedures . Enhanced Recovery After Surgery (ERAS) protocols offer a promising approach to optimize outcomes in this population.

Originally developed for colorectal surgery, ERAS principles have been successfully adapted to obstetric practice over the past decade. These evidence-based protocols emphasize multimodal interventions including preoperative counseling, optimized analgesia, early mobilization, and timely nutrition. In obstetrics, ERAS implementation has demonstrated reduced length of stay, decreased opioid use, and improved patient satisfaction for elective CS .

Application of ERAS to emergency CS requires special considerations due to the urgent nature of the procedure. Modified protocols focus on rapid preoperative assessment, regional anesthesia with intrathecal opioids, and immediate postoperative care initiation . Emerging evidence suggests these adaptations maintain benefits while accommodating time constraints . Key outcomes include reduced postoperative pain, earlier return of bowel function, and improved breastfeeding rates .

Current research demonstrates ERAS protocols can be safely implemented in emergency CS with proper staff training and institutional support . Ongoing studies continue to refine optimal practices, particularly regarding fluid management and thromboprophylaxis . As evidence accumulates, standardized guidelines for emergency CS ERAS pathways are expected to emerge .

DETAILED DESCRIPTION:
The study is conducted on two phases. First phase study tools will be prepared. This is followed by the first and second audit cycles, preparatory phase is done to assess the intra-operative and post-operative care of women undergoing emergency cesarean section using the guidelines of Enhanced recovery after Surgery society. The quality of recovery score-11 translated into arabic. Permission is sought from adminstritive authorities.

First audit cycle : compliance with intraoperative measures is obtained by direct observation . post-operative information will be obtained by patient interview and record audit. The quiality of recovery will be assessed just before discharge using the quality of recovery score (ObsQoR-11).

Corrective action : gaps identified by first audit cycle is translated into defined corrrective measures.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy who undergoing emergency cesarean section after 34weeks and accepting to be included in the study.

Exclusion Criteria:

* Pregnant woman who had previous rupture uterus.
* Other medical disorders as hypertensive disorder during pregnancy, cardiac disease.
* Intra-operative complications necessitating changes in post-operative care e.g. bowel injury, urinary tract injury.
* Hemodynamically unstable (post-partum hemorrhage)

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant patients admitted to Woman's Health hospital, Assiut university labor ward and post-partum.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
assess the obstetric ObQOR11scrore at 12 hours and 24 hours post-operative | From enrollment till discharge after 24 hours.
  A data collection tool will be prepared for the study. After screening for eligibility, demographic factors, obstetric history. weight and gain, quality of previous cesarean scar if any, hemoglobin will be assessed for all patients. Observation of the outcomes will be recorded in the first phase of the study using a structured proforma and the Arabic version of ObQOR-11 score. Secondary outcomes measures include first oral intake, first abulation, first urination after catheter removal, passage of flatus and pain visual analog scale every 4 hours till discharge.

SECONDARY OUTCOMES:
Secondary outcome | During hospital stay up to discharge, typically within 24-48 hours postoperative
  Time to first oral intake
Secondary outcome | During hospital stay up to discharge, typically within 24-48 hours postoperative
  Time to passage of flatus
Secondary outcome | During hospital stay up to discharge, typically within 24-48 hours postoperative
  Time to first ambulation
Secondary outcome | During hospital stay up to discharge, typically within 24-48 hours postoperative
  Time to first urination after catheter removal
Secondary outcome | During hospital stay up to discharge, typically within 24-48 hours postoperative
  Pain visual analog scale (VAS) scores every 4 hours until discharge